CLINICAL TRIAL: NCT03585452
Title: Effects of Dexmedetomidine on Cognitive Outcome and Brain Injury Markers After General Anesthesia for Cardiac Surgery on Cardiopulmonary Bypass
Brief Title: Effects of Dexmedetomidine on Cognitive Outcome and Brain Injury Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michał Kowalczyk (Other)
Responsible Party: Sponsor-Investigator, Michał Kowalczyk, Principal Investigator, Medical University of Lublin
Organization: Medical University of Lublin (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Cardiodex
Record Dates: First submitted 2018-07-01; First posted 2018-07-13 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cognitive Dysfunction
Keywords: dexmedetomidine; cardiac surgery; brain injury biomarkers; cognitive examination
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into two groups by simple 1:1 randomisation using opaque envelopes: the control group (group CON; patients with typical anaesthetic regimens) and the dexmedetomidine group (group DEX; those with additional dexmedetomidine infusion).
Who Masked: Participant
Masking Description: Patients were not aware of the fact into which group they were divided
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Active Comparator): Patients with typical anesthetic regimen: premedication: 2 mg estazolam p.o. and 10 mg morphine s.c. - 1 hour before procedure. Preoxygenation and induction of anaesthesia: remifentanyl 1 µg/kg, etomidate 0.3 mg/kg, pancuronium 0.1 mg/kg and intubation. Maintenance of the anesthesia: remifentanyl 0.2-0.5 µg/kg/min and propofol 2-4 mg/kg/min infusions. Ventilation with Air/O2. Additionally: nitroglycerine infusion or phenylephrine 0.05-0.1 mg boluses will be used for normotension maintenance at demanding doses. Subsequently typical CABG procedure with normothermic CPB will be performed. Weaning from CPB will be performed with inotropic support (dobutamine) and vasodilator (nitroglycerine) administration - with patients dependent doses. Routine recovery after surgery.
  Interventions: Drug: Propofol based general anesthesia
- Group D (Experimental): Regimen will be the same with additional dexmedetomidine infusion: with loading dose: 0.5 µg/kg/h through 1 hour and then dose will be reduced to 0.25 µg/kg/h and infusion will be continued during surgery and postoperative period to the total dose of 200 µg. Anesthetics and opioids doses will be adjusted under hemodynamic and eeg sensor - SedLine Masimo.
  Interventions: Drug: Dexmedetomidine Infusion

INTERVENTIONS:
Drug: Dexmedetomidine Infusion — Patients with additional dexmedetomidine infusion
  Other Names: Dexdor
  Arms: Group D
Drug: Propofol based general anesthesia — Patients with typical anaesthetic regimens
  Other Names: Control
  Arms: Group C

SUMMARY:
Dexmedetomidine is a drug with sedative, anxiolytic, and analgesic properties. Benefits of its use covers good sedations without respiratory suppression, reduced circulating catecholamines due to decreased sympathetic transmission and nociceptive transmission blocking resulting in lower needs for postoperative pain management. All these features are beneficial for cardiac surgery patients. What is more, it was find as an anesthesia agent.

Recently some protective effects were find, like reduced postoperative delirium occurrence with cardiac surgery dexmedetomidine sedated patients. Other study revealed that patient receiving dexmedetomidine during cardiac surgery and in the first 24 h postoperatively showed significant reductions in in-hospital and 30-day mortality as well as postsurgical delirium.

Although dexmedetomidine appears to reduce postoperative delirium, its role in prevention of neurological injury has not been well studied. To fulfil this gap we designed the study to investigate effects of dexmedetomidine use during cardiac surgery (with cardiopulmonary bypass - CPB) and in the first hours postoperatively on biomarkers of brain injury and cognitive function.

DETAILED DESCRIPTION:
All adult patients qualified for elective coronary artery bypass grafts (CABG), (with CPB), under general anesthesia with good ejection fraction - above 40% will be eligible for the study. Patients will be sampling by simple 1:1 sampling into 2 groups:

1. Control group (group C): patients with typical anesthetic regimen.
2. Dexmedetomidine group (group D): regimen will be the same with additional dexmedetomidine infusion.

In both groups typical monitoring will be applied: heart rate (HR), mean arterial pressure (MAP), systolic arterial pressure (SAP), diastolic arterial pressure (DAP), pulse oximetry (SpO2), central vein pressure (CVP), hemodynamic monitoring with Swan-Ganz thermodilution pulmonary artery catheter, end tidal carbon dioxide (ET CO2), typical inhaust and exhaust gases analysis, eeg sensor - SedLine with patient state index (PSI), (Masimo technology) and regional cerebral oximetry (Masimo technology) with estimation of area under curve defined as time of the low brain oximetry value below 80% of initial value.

Blood for bio-markers analysis will be collected in the following points:

1. initially, before anesthesia induction
2. At the end of the procedure
3. 24 hours after procedure
4. 72 hours after procedure Biochemical measures will cover: biomarkers of brain injury: myelin basic protein (MBP) and matrix metalloproteinase 12 (MMP12).

Cognitive function will be assessed using Addenbrooke's Cognitive Examination - ACE-III, at three time points: initially, one day before surgery, at discharge time and 3 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients qualified for elective coronary artery bypass grafts (CABG), (with CPB) with good ejection fraction - above 40%.

Exclusion Criteria:

* diabetic patients, neurological diseases, any autoimmune diseases, any internal carotid or vertebral artery obstruction, myocardial infarction, ejection fraction < 40%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Cognitive function | at discharge - 7 days after surgery
  Cognitive function assessment with Addenbrooke's Cognitive Examination - ACE-III

CONTACTS AND LOCATIONS:
Overall Officials: Michał Kowalczyk, M.D., Ph.D., Principal Investigator — Medical University of Lublin, Poland
Locations (1):
- Michał Kowalczyk, Lublin, Lublin Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
We plan to attach row data as supplemental data during publishing process.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available after article publication.
Access Criteria: Available for everybody.

REFERENCES:
- [Background] McDonagh DL, Berger M, Mathew JP, Graffagnino C, Milano CA, Newman MF. Neurological complications of cardiac surgery. Lancet Neurol. 2014 May;13(5):490-502. doi: 10.1016/S1474-4422(14)70004-3. Epub 2014 Apr 2. PMID 24703207
- [Background] Brandao PG, Lobo FR, Ramin SL, Sakr Y, Machado MN, Lobo SM. Dexmedetomidine as an Anesthetic Adjuvant in Cardiac Surgery: a Cohort Study. Braz J Cardiovasc Surg. 2016 May-Jun;31(3):213-218. doi: 10.5935/1678-9741.20160043. PMID 27737403
- [Background] Chen S, Hua F, Lu J, Jiang Y, Tang Y, Tao L, Zou B, Wu Q. Effect of dexmedetomidine on myocardial ischemia-reperfusion injury. Int J Clin Exp Med. 2015 Nov 15;8(11):21166-72. eCollection 2015. PMID 26885050
- [Background] Cheng H, Li Z, Young N, Boyd D, Atkins Z, Ji F, Liu H. The Effect of Dexmedetomidine on Outcomes of Cardiac Surgery in Elderly Patients. J Cardiothorac Vasc Anesth. 2016 Dec;30(6):1502-1508. doi: 10.1053/j.jvca.2016.02.026. Epub 2016 Mar 3. PMID 27435836
- [Background] Gong Z, Ma L, Zhong YL, Li J, Lv J, Xie YB. Myocardial protective effects of dexmedetomidine in patients undergoing cardiac surgery: A meta-analysis and systematic review. Exp Ther Med. 2017 May;13(5):2355-2361. doi: 10.3892/etm.2017.4227. Epub 2017 Mar 13. PMID 28565849
- [Background] Ji F, Li Z, Young N, Moore P, Liu H. Perioperative dexmedetomidine improves mortality in patients undergoing coronary artery bypass surgery. J Cardiothorac Vasc Anesth. 2014 Apr;28(2):267-73. doi: 10.1053/j.jvca.2013.06.022. Epub 2013 Oct 29. PMID 24182835
- [Background] Perez-Zoghbi JF, Zhu W, Grafe MR, Brambrink AM. Dexmedetomidine-mediated neuroprotection against sevoflurane-induced neurotoxicity extends to several brain regions in neonatal rats. Br J Anaesth. 2017 Sep 1;119(3):506-516. doi: 10.1093/bja/aex222. PMID 28969317
- [Background] Wang Y, Han R, Zuo Z. Dexmedetomidine-induced neuroprotection: is it translational? Transl Perioper Pain Med. 2016;1(4):15-19. PMID 28217717
- [Background] van Dijk D, Keizer AM, Diephuis JC, Durand C, Vos LJ, Hijman R. Neurocognitive dysfunction after coronary artery bypass surgery: a systematic review. J Thorac Cardiovasc Surg. 2000 Oct;120(4):632-9. doi: 10.1067/mtc.2000.108901. PMID 11003741
- [Background] Mioshi E, Dawson K, Mitchell J, Arnold R, Hodges JR. The Addenbrooke's Cognitive Examination Revised (ACE-R): a brief cognitive test battery for dementia screening. Int J Geriatr Psychiatry. 2006 Nov;21(11):1078-85. doi: 10.1002/gps.1610. PMID 16977673
- [Background] Ottens AK, Golden EC, Bustamante L, Hayes RL, Denslow ND, Wang KK. Proteolysis of multiple myelin basic protein isoforms after neurotrauma: characterization by mass spectrometry. J Neurochem. 2008 Mar;104(5):1404-14. doi: 10.1111/j.1471-4159.2007.05086.x. Epub 2007 Nov 22. PMID 18036155
- [Background] Chelluboina B, Warhekar A, Dillard M, Klopfenstein JD, Pinson DM, Wang DZ, Veeravalli KK. Post-transcriptional inactivation of matrix metalloproteinase-12 after focal cerebral ischemia attenuates brain damage. Sci Rep. 2015 May 8;5:9504. doi: 10.1038/srep09504. PMID 25955565